CLINICAL TRIAL: NCT03943407
Title: Characterization of the Toll-like Receptor 7-agonist Imiquimod 3.75% As a New Surrogate Model of Itch
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Imiquimod 3.75% was ineffective
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190029
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2021-01

CONDITIONS: Itch
Keywords: Imiquimod; Doxepin; Trans-cinnamaldehyde (CA); L-menthol; Histamine; Cowhage
MeSH Terms: conditions — Pruritus | interventions — Imiquimod; Doxepin; Histamine; Menthol; cinnamaldehyde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Zyclara/vehicle (Experimental): All subjects will be treated with Zyclara cream (Imiquimod 3.75%) and vehicle.
  Interventions: Drug: Zyclara 3.75 % Topical Cream
- Zyclara/Doxepin (Experimental): All subjects will be treated with the topical antihistamine cream (Prudoxin, containing 5% doxepin hydrochloride, Healthpoint, San Antonio, TX) or a placebo cream. After removal, subjects will be treated with Zyclara cream
  Interventions: Drug: Zyclara 3.75 % Topical Cream; Drug: Prudoxin
- Zyclara/Histamine/Cowage (Experimental): All subjects will be treated with Zyclara cream, vehicle cream, histamine and cowhage
  Interventions: Drug: Zyclara 3.75 % Topical Cream; Other: Histamine; Other: Cowhage
- Zyclara/L-menthol/trans-cinnamaldehyde (Experimental): All subjects will be treated with Zyclara cream (Imiquimod 3.75%) and vehicle. After removal, subjects will be treated with L/menthol and trans-cinnamaldehyde
  Interventions: Drug: Zyclara 3.75 % Topical Cream; Other: L-menthol; Other: Trans-cinnamaldehyde (CA)

INTERVENTIONS:
Drug: Zyclara 3.75 % Topical Cream — The cream will be applied on 4x4 cm squared areas on the volar forearm. The cream will be left in place for 2h, 1 h or 30 min (sub-study 1) after which it will be removed. The technical and security procedures will be conducted in accordance with the manufacturer's instructions.
Drug: Prudoxin — The anti-histamine cream Prudoxin, containing 5% doxepin hydrochloride (1 g contains 50 mg of doxepin) (Healthpoint, San Antonio, TX) will be applied on the volar forearm. Two adhesive patches 4×4 cm (1mm thick, 3M foam adhesive tape, 3M, St. Paul, MN) each with a 3.5×3.5 cm center cut out (to deposit 1.2 grams of cream) will be each placed 3 cm distal and 3 cm proximal to the center of the volar aspect of each arm. Each patch will be covered with Tegaderm I.V., an occlusive, adhesive dressing (3M), for at least 1 h and 30 minutes.
  Arms: Zyclara/Doxepin
Other: Histamine — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied. The lancets have a 1 mm shouldered tip adapt to introduce a small amount of test substance extremely locally and approximately at the dermo-epidermal junction. . A small drop of histamine dihydrochloride (1%, in saline) will be applied to a previously determined area on the volar forearm followed by a prick through the drop.
  Arms: Zyclara/Histamine/Cowage
Other: Cowhage — Cowhage spicules are 1-2 mm in length and have diameter of 1-3 um at their tip. The active substance delivered (mucunain) has been calculated to be in the nanogram range. The insertion of cowhage spicule(s) rapidly and consistently produces itch with no or very little flare reaction. This insertion is conducted by forceps using a stereo-microscope, and 30-35 spicules are gently rubbed into a 1 cm diameter skin area.
  Arms: Zyclara/Histamine/Cowage
Other: L-menthol — L-menthol (≥99.9%, TRPM8 agonist; (Sigma Aldrich, Broendby, Denmark) is dissolved in 96% ethanol at concentrations of 40%(w/v) L-menthol. A 1 mL aliquot is dispensed onto a 3 × 3 cm cotton pad and placed on a 6 × 6 cm sheet of medical tape. In between the cotton pad and the medical tape, a layer of parafilm will be added to avoid evaporation. This configuration was subsequently applied for 1 h.
  Arms: Zyclara/L-menthol/trans-cinnamaldehyde
Other: Trans-cinnamaldehyde (CA) — CA will be obtained from Sigma Aldrich (Brøndby, Denmark) and dissolved in 90% ethanol at a concentration of 10% (vol/vol) CA. One ml aliquot of CA is dispensed onto a 3x3 cm cotton pad and placed on a 5x5 cm sheet of medical tape. Between the cotton pad and the tape, a layer of plastic film will be added to inhibit the evaporation of the solutions. This configuration will be applied for 1 h.
  Arms: Zyclara/L-menthol/trans-cinnamaldehyde

SUMMARY:
The aim of this research project is to design a new model of human itch by application of Zyclara cream. Further, the aim is to characterize the model and to verify if the mechanism of action of imiquimod follows the histaminergic or non-histaminergic pathway by using the anti-histamine drug doxepin. The last goal is to evaluate the interaction between the activation of TLR7 receptor and the activation of TRPA1 and TRPM8 receptors, which are two of the most important receptors involved in the transduction of noxious stimuli, and to evaluate to which extent these three channel populations functionally overlap.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Superficial blood perfusion by by a Speckle contrast imager (FLPI, Moor Instruments, England). | Change from baseline, to maximum 19 days after intervention
  Two pictures will be taken: one with the sensor placed approximately 35 cm above the induction area and one with the sensor placed approximately 20 cm above the induction area.
Trans-epidermal Water Loss (TEWL) | Change from baseline, to maximum 19 days after intervention
  a 2x2 cm hollow probe with two small humidity gauges and two thermometers is placed lightly on the skin for 10-25 seconds. These establish a precise humidity gradient in a 2 cm vicinity of the skin, representative for the point-loss of water though the epidermis.
Neurogenic Inflammatory Response and Pigmentation | Change from baseline, to maximum 19 days after intervention
  treatment will be measured with a spectrometer designed for cutaneous use (ColorMeter, DSM II; Cortex Technology, Hadsund, Denmark).
Measuring Alloknesis | Change from baseline, to maximum 19 days after intervention
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Thermal measurements (cold and warm detection thresholds, cold and heat pain thresholds) | Change from baseline, to maximum 19 days after intervention
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Measurement of Pain to Supra-threshold Heat Stimuli | Change from baseline, to maximum 19 days after intervention
  The test will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Measurement of Mechanical Detection Thresholds, Mechanical Pain Threshold and sensitivity | Change from baseline, to maximum 19 days after intervention
  These tests are conducted using a set of 20 different von Frey hairs (North Coast Medical, Gilroy, CA) with exerted forces ranging from .008g to 300g.

SECONDARY OUTCOMES:
Measurement of Itch rating by Computerized Visual Analog Scale Scoring | Change from baseline, to maximum 19 days after intervention
  We will ask the subjects to rate the sensation of itch on a VAS scale ranging from 0 to 10 where 0 indicates "no itch" and 10 indicates "worst itch imaginable"to 10 where 0 indicates "no itch" and 10 indicates "worst itch imaginable" and similarly for sensations of stinging/pricking and burning, both of which are frequently associated with the sensation of itch or pain.
Measurement of pain rating by Computerized Visual Analog Scale Scoring | Change from baseline, to maximum 19 days after intervention
  the subjects will be asked to rate the sensation of pain on a VAS scale ranging from 0 to 10 where "0" is no pain and "10" is the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No